CLINICAL TRIAL: NCT00070876
Title: Trial of Psychosocial Training for Pediatric Generalists
Brief Title: Psychosocial Training for Pediatric Health Care Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lawrence Wissow, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: R01MH062469 (NIH); R01MH062469 (NIH); DSIR 82-SPEC
Record Dates: First submitted 2003-10-08; First posted 2003-10-09 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Mental Disorders Diagnosed in Childhood
Keywords: Child; Adolescent
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Mental health communication skills training

SUMMARY:
This study will provide psychosocial training to general health care providers to help them provide better care to children with mental health problems.

DETAILED DESCRIPTION:
Up to 20% of school-age children have one or more mental health conditions that require treatment. These conditions are often treated by generalists. However, a significant proportion of children who seek treatment from generalists do not receive effective treatment. Studies indicate that generalists who treat adults can improve the administration of treatment after taking part in training programs, but these studies have yet to be translated into pediatric settings. This study will conduct a training program to help generalists provide effective treatments to children with mental health problems.

This study will evaluate a two-session, highly interactive training program in which general clinicians receive psychosocial training. The training program includes skills related to engaging parents and children, problem identification, solution-focused cognitive therapy, and making effective mental health referrals.

The child's mental health symptoms, functioning, changes in utilization of pediatric services, and utilization of community services will be measured along with the mother's emotional well-being and family functioning.

ELIGIBILITY:
Inclusion Criteria for Health Care Providers:

* Generalist clinician in primary care practice seeing children 6 to 16 years of age

Inclusion Criteria for Patients:

* 6 to 16 years of age
* Seeing a study-enrolled provider
* English or Spanish speaking
* Not in acute pain

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350
Dates: Start 2002-08; Primary Completion 2005-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Wissow LS, Gadomski A, Roter D, Larson S, Brown J, Zachary C, Bartlett E, Horn I, Luo X, Wang MC. Improving child and parent mental health in primary care: a cluster-randomized trial of communication skills training. Pediatrics. 2008 Feb;121(2):266-75. doi: 10.1542/peds.2007-0418. PMID 18245417